CLINICAL TRIAL: NCT00349518
Title: A Phase II Study of Dasatinib (BMS-354825) in Subjects With Chronic or Advanced Phase Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Who Are Resistant or Intolerant to Imatinib
Brief Title: Study of Dasatinib in Imatinib Resistant or Intolerant Subjects With Chronic or Advanced Phase CML or Philadelphia Chromosome Positive ALL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-083; EUDRACTnr: 2006-001279-39
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Chronic and Advanced Phase CML and; Philadelphia Chromosome Positive ALL with imatinib intolerance or resistance
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Bronchiolitis Obliterans Syndrome | interventions — Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
The purpose of this study is to further assess the safety of dasatinib in imatinib intolerant or resistant patients with chronic phase chronic myeloid leukemia, advanced phase chronic myeloid leukemia or Philadelphia chromosome positive acute lymphoblastic leukemia. The efficacy of the drug in this kind of patients will also further be documented.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 or older
* CP or AD CML or Ph+ ALL
* Intolerant of resistant to imatinib
* ECOG PS 0-2 (CP CML)
* ECOG PS 0-3 (AD CML and Ph+ ALL)
* Adequate hepatic and renal function

Exclusion Criteria:

* Pregnant or breastfeeding females
* History of significant cardiac disease
* History of significant bleeding disorder (not CML)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of drug-related adverse events.

SECONDARY OUTCOMES:
Chronic Phase CML: Cytogenetic and Hematologic Response
Advanced Phase CML and Philadelphia positive ALL: Hematologic Response
Time to and duration of Cytogenetic and Hematologic Response

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- Local Institution, Budapest, Hungary
- Italy (3):
  - Local Institution, Bologna
  - Local Institution, Orbassano (To)
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Poland (6):
  - Local Institution, Gdansk
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Instiution, Lodz
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- United Kingdom (6):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Newcastle, Tyne and Wear
  - Local Institution, Birmingham, West Midlands